CLINICAL TRIAL: NCT00000800
Title: Methadone Effects on Zidovudine (ZDV, AZT) Disposition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 262; 11239 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Methadone; Drug Interactions; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Methadone; Zidovudine

INTERVENTIONS:
Drug: Methadone hydrochloride
Drug: Zidovudine

SUMMARY:
To determine whether methadone maintenance alters the pharmacokinetics of zidovudine (AZT). To determine whether any such effect of methadone on disposition of AZT is time dependent and whether a metabolic interaction between AZT and methadone exists.

Injection drug users represent an increasing proportion of HIV-infected persons. Since daily methadone maintenance is the major chemical treatment for injection drug abuse, it is important to determine the impact of methadone on AZT absorption, distribution, and elimination.

DETAILED DESCRIPTION:
Injection drug users represent an increasing proportion of HIV-infected persons. Since daily methadone maintenance is the major chemical treatment for injection drug abuse, it is important to determine the impact of methadone on AZT absorption, distribution, and elimination.

After 6 days of inpatient detoxification with clonidine, patients addicted to opiates are randomized to receive either oral or intravenous AZT for the first dose, followed by determination of plasma and urine pharmacokinetics. On the second day of AZT dosing, the alternate form of administration will be used for the first dose. On both days, all other doses are given orally. Patients then begin methadone maintenance in combination with AZT for 7 days of inpatient treatment, with further pharmacokinetic sampling. After hospitalization for 16 days total, patients continue AZT/methadone treatment on an outpatient basis, and then 2 months later are readmitted as inpatients for 5 days for further pharmacokinetic sampling. Control patients who are not addicted to opiates are hospitalized for 3 days at study entry and are randomized for AZT treatment and pharmacokinetic sampling in the same manner as the first group, although they will not receive methadone treatment. Control patients are readmitted for 2 days after 1 week of AZT treatment and then again after 59 days of AZT treatment.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 count 100 - 500 cells/mm3.
* No active opportunistic infection or wasting syndrome.
* Opiate addiction or prior enrollment in a methadone treatment program (methadone recipients only).
* Admission to General Clinical Research Center at Yale-New Haven Hospital for clonidine detoxification (methadone recipients only).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Inadequate IV access.
* Benzodiazepine abuse.

Concurrent Medication:

Excluded:

* Amiodarone.
* Anesthetics, general.
* Azithromycin.
* Barbiturates.
* Carbamazepine.
* Cimetidine.
* Ciprofloxacin.
* Clarithromycin.
* Dexamethasone.
* Disulfiram.
* Erythromycin.
* Fluoroquinolones.
* Fluoxetine.
* Gestodene.
* Hydrochlorothiazide.
* Hypoglycemics, oral.
* Isoniazid.
* Itraconazole.
* Ketoconazole.
* Levomepromazine.
* MAO inhibitors.
* Methoxsalen.
* Nafcillin.
* Narcotic analgesics.
* Naringenin.
* Norethindrone.
* Omeprazole.
* Pentazocine.
* Phenothiazines.
* Phenytoin.
* Quinidine.
* Ranitidine.
* Rifabutin.
* Rifampin.
* Sedative Hypnotics.
* Sulfaphenazole.
* Tranquilizers (except at discretion of investigator and protocol chair).
* Tricyclic antidepressants.
* Troleandomycin.
* Warfarin.

Prior Medication:

Excluded within 4 weeks prior to study entry:

* Rifampin or its derivatives.
* Phenytoin.
* Barbiturates.
* Cimetidine.
* Other drugs known to induce or inhibit hepatic microsomal enzymes.

Excluded within 14 days prior to study entry:

* Any other experimental drug.
* Drugs with known nephrotoxic potential.

Excluded within 72 hours prior to study entry:

* Amiodarone.
* Anesthetics, general.
* Azithromycin.
* Carbamazepine.
* Ciprofloxacin.
* Clarithromycin.
* Dexamethasone.
* Disulfiram.
* Erythromycin.
* Fluoroquinolones.
* Fluoxetine.
* Gestodene.
* Hydrochlorothiazide.
* Hypoglycemics, oral.
* Isoniazid.
* Itraconazole.
* Ketoconazole.
* Levomepromazine.
* MAO inhibitors.
* Methoxsalen.
* Nafcillin.
* Narcotic analgesics.
* Naringenin.
* Norethindrone.
* Omeprazole.
* Pentazocine.
* Phenothiazines.
* Quinidine.
* Ranitidine.
* Rifabutin.
* Sedative Hypnotics.
* Sulfaphenazole.
* Tranquilizers (except at discretion of investigator and protocol chair).
* Tricyclic antidepressants.
* Troleandomycin.
* Warfarin.

Continued active drug or alcohol abuse or dependence that would decrease the probability of study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jatlow P, Study Chair; Rainey P, Study Chair
Locations (1):
- Yale Univ / New Haven, New Haven, Connecticut, United States

REFERENCES:
- [Background] Jatlow P, Mccance EF, Rainey PM, Trapnell CB, Friedland G. Methadone increases zidovudine exposure in HIV-infected injection drug users (ACTG 262). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:129
- [Background] McCance-Katz EF, Rainey PM, Jatlow P, Friedland G. Methadone effects on zidovudine disposition (AIDS Clinical Trials Group 262). J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Aug 15;18(5):435-43. doi: 10.1097/00042560-199808150-00004. PMID 9715839